CLINICAL TRIAL: NCT03482713
Title: Phase II Study, Randomized, Double-Blind, Placebo-Controlled 4-Week Clinical Study, to Evaluate the Efficacy and Safety of MK-7264 in Adult Japanese Participants With Unexplained or Refractory Chronic Cough
Brief Title: Study of Gefapixant (MK-7264) in Adult Japanese Participants With Unexplained or Refractory Chronic Cough (MK-7264-033)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-033; MK-7264-033 (Other: Merck Protocol Number); 183925 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Intervention Model Description: Japanese adult participants with refractory or unexplained chronic cough will be randomized to 1 of 2 treatment groups: gefapixant 45 mg twice daily (BID), or placebo BID.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gefapixant 45 mg (Experimental): Participants will receive a gefapixant 45 mg film-coated tablet BID for 28 days.
  Interventions: Drug: Gefapixant 45 mg
- Placebo (Placebo Comparator): Participants will receive a film-coated placebo tablet matching gefapixant BID for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant 45 mg — Gefapixant 45 mg (film-coated tablet) to be administered orally BID
  Other Names: MK-7264
  Arms: Gefapixant 45 mg
Drug: Placebo — Placebo (film-coated tablet) matching gefapixant to be administered orally BID
  Arms: Placebo

SUMMARY:
This estimation study (no hypotheses) will evaluate the safety, tolerability, and efficacy of gefapixant (MK-7264) in Japanese adult participants with unexplained or refractory chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography scan of the thorax (within 5 years of Screening/Visit 1 and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease in the opinion of the principal investigator or the sub-investigator.
* Has had chronic cough for ≥ 1 year and a diagnosis of refractory chronic cough or unexplained chronic cough.
* For female participants, is a female who is not pregnant, not breastfeeding, not of childbearing potential, or agrees to follow contraceptive guidance
* Provides written informed consent and is willing and able to comply with the study protocol (including use of the digital cough recording device and completion of study questionnaires)

Exclusion Criteria:

* Is a current smoker or has given up smoking within 12 months of Screening, or is a former smoker with a pack-year history >20 pack-years
* Has a history of upper or lower respiratory tract infection or recent clinically significant change in pulmonary status
* Has a history of chronic bronchitis
* Is currently taking an angiotensin converting enzyme inhibitor (ACEI), or has used an ACEI within 3 months of Screening
* Has a history of malignancy ≤5 years
* Has a screening systolic blood pressure >160 millimeters of mercury (mmHg) or a diastolic blood pressure >90 mm Hg
* Has a history of cutaneous adverse drug reaction to sulfonamides with or without systemic symptoms or history of anaphylaxis to sulfonamides
* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence
* Has a known allergy/sensitivity or contraindication to gefapixant
* Has donated or lost ≥1 unit of blood within 8 weeks prior to the first dose of gefapixant
* Has previously received gefapixant or is currently participating in or has participated in an interventional clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- Japan (16):
  - Nagoya City University Hospital ( Site 3328), Nagoya, Aichi-ken
  - Idaimae Minamiyojo Int Clinic ( Site 3321), Sapporo, Hokkaido
  - Tsumura Cardiovascular-internal-medicine Clinic ( Site 3314), Kakogawa, Hyōgo
  - Hitachi, Ltd. Hitachinaka General Hospital ( Site 3301), Hitachi-Naka, Ibaraki
  - Saiseikai Kanazawa Hospital ( Site 3337), Kanazawa, Ishikawa-ken
  - Komatsu Municipal Hospital ( Site 3308), Komatsu, Ishikawa-ken
  - Kamei Internal Medicine and Respiratory Clinic ( Site 3309), Takamatsu, Kagawa-ken
  - Yokohama City Minato Red Cross Hospital ( Site 3306), Yokohama, Kanagawa
  - Matsusaka City Hospital ( Site 3325), Matsusaka, Mie-ken
  - Nagaoka Red Cross Hospital ( Site 3307), Nagaoka, Niigata
  - Kawaguchi Respiratory Clinic ( Site 3304), Higashiosaka, Osaka
  - Fukushima Medical University Hospital ( Site 3338), Fukushima
  - Doujin Memorial Medical Foundation, Meiwa Hospital ( Site 3310), Tokyo
  - Nihonbashi Medical & Allergy Clinic ( Site 3334), Tokyo
  - Fukuwa Clinic ( Site 3311), Tokyo
  - Showa University Hospital ( Site 3331), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefapixant 45 mg: Participants received a gefapixant 45 mg film-coated tablet twice daily for 28 days.
- Placebo: Participants received a film-coated placebo tablet matching gefapixant twice daily for 28 days.
Period: Overall Study
Arm/Group | Gefapixant 45 mg | Placebo
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant 45 mg | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (15.7) | 57.2 (11.7) | 55.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 11 | 12 | 23
24-hour cough frequency [Mean (Standard Deviation); unit: coughs/hour] | 40.1 (86.7) | 22.9 (20.5) | 31.1 (60.9)
Awake cough frequency [Mean (Standard Deviation); unit: coughs/hour] | 49.0 (103.0) | 27.3 (21.0) | 37.7 (71.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 6 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant 45 mg | Placebo
Number analyzed (Participants) | 11 | 12
Participants | 9 | 2

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to 4 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant 45 mg | Placebo
Number analyzed (Participants) | 11 | 12
Participants | 1 | 0

3. Secondary Outcome: Change From Baseline at Week 4 in Log-transformed 24-hour Coughs Per Hour
Description: Cough frequency will be evaluated using a digital recording device which records sounds from the lungs and trachea through a chest contact sensor, as well as ambient sounds through a lapel microphone. Change from baseline in log-transformed 24-hour coughs per hour = log (24-hour coughs per hour at post-baseline) - log (24-hour coughs per hour at baseline). The denominators may be different if the recording period is actually <24 hours but ≥20 hours).
Time Frame: Baseline and Week 4
Population: All randomized participants who have taken at least one dose of study medication and provided at least one baseline and one post-baseline 24-hour cough observations during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant 45 mg | Placebo
Number analyzed (Participants) | 11 | 12
Coughs/hour | -0.23 (0.39) | -1.02 (0.38)
Statistical Analysis 1: Comparison: Gefapixant 45 mg vs Placebo; Test type: Other; Difference in least squares means = 0.79, 95% CI 2-sided [-0.34 to 1.93] — Based on an ANCOVA model with terms for treatment, gender and the log-transformed baseline

4. Secondary Outcome: Change From Baseline at Week 4 in Log-transformed Awake Coughs Per Hour
Description: Change from baseline at Week 4 in awake coughs per hour is the average hourly cough frequency (based on sound recordings) during the 24-hour monitoring period while the participant is awake. Change from baseline in log-transformed awake coughs per hour = log (awake coughs per hour at post-baseline) - log (awake coughs per hour at baseline) for the monitoring period the participant is awake.
Time Frame: Baseline and Week 4
Population: All randomized participants who have taken at least one dose of study medication and provided at least one baseline and one post-baseline awake cough observations during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: Coughs/hour
Arm/Group | Gefapixant 45 mg | Placebo
Number analyzed (Participants) | 11 | 12
Coughs/hour | -0.20 (0.38) | -0.97 (0.37)
Statistical Analysis 1: Comparison: Gefapixant 45 mg vs Placebo; Test type: Other; Difference least squares mean = 0.76, 95% CI 2-sided [-0.35 to 1.88] — Based on an ANCOVA model with terms for treatment, gender and the log-transformed baseline

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Gefapixant 45 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 9/11 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 45 mg (N=11) | Placebo (N=12)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 7 (7) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03482713/Prot_SAP_000.pdf